Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

#### **KEY INFORMATION FOR**

# PRAGMATIC, RANDOMIZED, BLINDED TRIAL TO SHORTEN PHARMACOLOGIC TREATMENT OF NEWBORNS WITH NEONATAL OPIOID WITHDRAWAL SYNDROME (NOWS) INFORMED CONSENT FORM FOR BABY ONLY

NOTE: "You" and "your baby" refer to the caregiver - be that biological parent or other legal guardian.

We are asking you to choose whether or not you want your baby to participate in a clinical trial (research study) about babies who have neonatal opioid withdrawal syndrome (NOWS). Neonatal opioid withdrawal syndrome can cause a number of problems. These problems may include tremors, seizures, fussiness, vomiting, and poor feeding. Babies can develop NOWS if their mothers took drugs called opioids while the babies were still inside their mothers. There are many different names for opioids. Some brand names, generic names, and street names are listed on the last page of this form.

# **Before delivery:**

Because your baby may have been exposed to opioids during pregnancy, your baby could have NOWS after he/she is born. If your baby does have NOWS after he/she is born, your baby's doctor and medical team will help him/her to get over it. The doctor may give him/her a drug (either morphine or methadone) that will help your baby get over NOWS.

#### After delivery:

Your baby has or may have NOWS and is currently being given a drug (either morphine or methadone) by his/her doctor to help him or her get over NOWS.

Your baby will need to be weaned (slowly stop getting) from the drug so that your baby will get better. The question the researchers want to answer is whether or not there is a difference between a slow weaning method and a fast weaning method.

This page and the next 2 pages give you key information to help you decide whether to allow your baby to participate. We have included detailed information after the third page. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is below.

#### WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

By doing this study, we hope to learn about the best way babies can stop getting the morphine or methadone the doctors may be using to treat your baby if your baby has NOWS symptoms.

Informed Consent BABY ONLY Template Version #: 03 cIRB# 260053
Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

If your baby needs medicine to help with the NOWS symptoms while he/she is in the hospital, and if you agree to volunteer for this study, your baby will be placed in one of two groups, "slow weaning" or "fast weaning." If your baby does not need medicine for NOWS symptoms, we will let you know and your baby will not stay in the study.

In some hospitals, doctors use a SLOW WEANING approach, in which the baby spends more time on morphine or methadone, and in other hospitals doctors use a FAST WEANING approach, in which the baby spends less time on morphine or methadone. Nobody knows which approach is better for the baby. The question the researchers want to answer is whether one of these 2 approaches is better than the other. Details about these groups are given in the section "What will happen if I say yes, I want my baby to be in this study?" in the main part of the consent form. During your baby's hospital stay, medical and research staff will complete the weaning process, collect information about what medicines are used and how much is given, The staff will also track your baby's health. The research team will check your baby's size and weight when your baby is ready to leave the hospital. After your baby leaves the hospital the research team will ask you to answer questionnaires that will occur via phone, electronically, or in person. These questionnaires ask about how well you and your baby are doing and will ask you to bring your baby in for tests on how well he/she is developing. The questionnaires will include things like how your baby is feeding, how your baby behaves, and about any urgent care hospital visits for your baby after your baby is home. You will be asked to bring your baby in for a play-based exam that will allow medical professionals to determine how well your child is developing compared to other babies his/her age.

Your and your baby's participation in this research will take about 4 hours over the course of about 2 years after your baby has been discharged from the hospital. The length of the hospital portion will depend on your baby's responses to the treatment, but is likely to be less than 30 days. There will be a total of 6 contact times. The first (at discharge) and last (when your baby is 24-months old) will be in person. The other 4 times will be either phone calls, home visits, or be done electronically.

#### WHY MIGHT I CHOOSE TO VOLUNTEER FOR THIS STUDY?

Your baby may not benefit directly from being in this study. Although there is no guarantee your baby will benefit directly, benefits could include one or more of the following:

less exposure to morphine or methadone

For a complete description of benefits, refer to the Full Consent.

#### WHY MIGHT I CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

The reason(s) you may not want your baby to be a volunteer for this study include:

- You might be uncomfortable sharing private health information about your baby with the research team.
- Fast weaning (versus slow weaning) could increase signs of NOWS for your baby.

Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

 It is possible that slow weaning could result in your baby receiving more days of morphine or methadone than with fast weaning.

For a complete description of risks, refer to the Full Consent.

If you chose not to have your baby be part of this study, your baby's treatment will be the hospital's usual care, which will be treatment with either morphine or methadone and changes in dose will be made by your baby's medical team. For a complete description of alternate treatment/procedures, refer to the Full Consent and/or ask your doctor.

#### DO I HAVE TO TAKE PART IN THE STUDY?

No. It is okay to say no. If you decide to take part in the study and let your baby be in the study, it should be because you really want to volunteer for your baby. You/your baby will not lose any services, benefits, or rights you/your baby would normally have if you choose not to volunteer for your baby.

If you want to know more about the research, let the study team know so they can give you more information.

Also tell the study team if you have decided you don't want to be in the study. It is perfectly okay to say no.

Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

# <Insert local institution name>

# **Informed Consent Form**

- We are asking you to allow your baby to be in a clinical trial (research study). You do not have to allow your baby to join the study.
- You/your baby will still get medical care from [insert local context here] even if your baby is not in the study.
- Please take as much time as you need to read this form and decide what is right for vou/vour baby.

In this consent form, the terms "I" refers to both you/ your baby.

# Why am I being asked to allow my baby to be in this clinical trial (research study)?

- We want to learn more about how to help babies born with Neonatal Opioid Withdrawal Syndrome (NOWS). Babies who, while growing inside their mothers, have been exposed to opioids can have NOWS. There are many names for opioids. Some of the brand names, generic names, and street names are listed on the last page of this form. The signs of NOWS are different in different babies. Signs can include tremors, seizures, fussiness, vomiting, poor feeding, as well as many other symptoms.
- This study may help us learn more about which method(s) might work better than others for treating NOWS. Specifically, the research team is testing whether it may be better to wean babies fast or slow from the methadone or morphine that is being used to treat babies' NOWS symptoms.
- We are asking people like you/your baby, who may have NOWS, to help us.
- Approximately 502 babies who are being treated with methadone or morphine for NOWS will be in this study. The babies' parent/legal guardian will also be in the study, if they want to be.
- This clinical trial (research study) is sponsored by the National Institutes of Health and is being conducted at about 24 hospitals across the United States.

#### What if I don't understand something?

• This form may have words you don't understand. If you'd like, research staff will read and explain it with you.

Informed Consent BABY ONLY Template Version #: 03

Template Date: 28-July-2021


Study Title: Pragmatic, Randomized, Blinded Trial to Shorten Pharmacologic Treatment of Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

- You are free to ask questions at any time before, during, or after your baby is in the study.
- Please ask as many questions as you like before you decide whether you want to allow your baby to be in this study.

# What will happen if I say yes, I want my baby to be in this study?

We first will see if your baby qualifies to be in the study. We will make sure that your baby

- Was inside his/her mother for at least 36 weeks.
- Is at risk for having NOWS or is receiving morphine or methadone to treat NOWS but weaning has not started.
- Can receive medicines by mouth or by nasogastric tube.
- Is being fed by mouth.

Your baby can not be part of this study if he or she has (or had) certain medical problems. The person who is going over this consent with you can list these problems if you want to know what they are.

If you want your baby to be in this study, we will do these things:

- Ask you to sign this consent form.
- We will monitor your baby for signs of NOWS to see if he/she qualifies to be in the study.
- If your doctors have started giving your baby morphine or methadone to treat NOWS, we will make sure he/she is on a stable amount. We will also make sure the doctors have not started reducing the amount yet.
- Let you know if your baby does not qualify to be in the study.
- The amount (dose) of morphine or methadone your baby will receive will be lowered in steps. If your baby is showing signs that he/she is having problems with the lowered amount, the amount will be raised to help your baby.
- Tell you that your baby will be placed in 1 of 2 different groups. Your baby will continue to receive the medication that her or his doctor is currently prescribing (morphine or methadone). However, the steps used to decrease the dose in group 1 will be different than the steps used to decrease the dose in group 2. One group will have medication decreased faster than the other group. The chances your baby will be in either group is the same as flipping a coin and getting either heads or tails. You will not know if your baby was put in the fast weaning or slow weaning group. Your doctor and nurses will not know if your baby was put in the fast weaning or slow weaning group. However, we can find out which group your baby is in if we need to in an emergency.

Informed Consent BABY ONLY Template Version #: 03

Template Date: 28-July-2021


Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

- Babies in both groups will go through 8 steps of study drug. Babies in the slow weaning group will have the dose of the drug decreased in 8 steps. Babies in the fast weaning group will have the dose decreased in 5 steps, and then they will receive a placebo (no medicine, like salt water) for 3 steps. The steps will be changed based on how your baby is doing and his or her needs. The amount of time your baby is in the hospital will be the same no matter which group your baby is assigned to.
- Your baby will continue to get morphine or methadone until he or she is stable without either morphine or methadone.
- The length of time your baby is in this study will depend on how he/she responds to the lowering of the amount of morphine or methadone.
- We will assess your baby's well-being using questionnaires. Questionnaires will be done electronically, over the phone, or in person. You do not have to answer any questions you do not want to answer. The description and schedule for these questionnaires are listed in the "Contact Times" below.
- We will assess your child's behavior and development. This will be done on your baby 24 to 48 hours after your baby has stopped getting methadone or morphine. This will help the medical team evaluate your baby's behavior. The assessment includes determining how calm or excitable the baby is, how well she or he takes to being handled, and how easily he or she can be made more comfortable. This is a physical exam. It involves moving your baby's arms and legs and watching the baby closely.
- Your baby will be watched in the hospital for 48 to 72 hours after he/she stops getting study drug. The medical team will watch closely for any signs of NOWS. If your baby still needs the study drug, it can be restarted.
- During your baby's hospital stay, you/your baby will receive your hospital's usual care except for the following:
  - ✓ Your baby's medical team will not decide how fast or slow your baby is weaned from methadone or morphine. Instead, your baby will be randomly put into either the "fast weaning group" or the "slow weaning group." The chance of your baby being in either group is like the chance of getting heads or tails when you flip a coin. The chance your baby will be into the fast weaning group is exactly the same as the chance your baby will be put into the slow weaning group.
  - ✓ Your baby will be assessed for nervous system, behavioral, and motor development.
  - ✓ Collection of information about your baby when your baby is discharged from the hospital. This information will be from the hospital records of your baby's biological mother and of your baby and will include things like your baby's size and weight and medication(s) used.

Template Date: 28-July-2021 

Study Title: Pragmatic, Randomized, Blinded Trial to Shorten Pharmacologic Treatment of Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

# Description of Post-Discharge Assessments

- You will be asked to provide contact information.
- You will be asked to answer questionnaires about how your baby is feeding and about any urgent care/emergency room visits or hospitalization that happened after your baby was sent home.
- You will be asked to bring your baby in so a medical professional can:
  - ✓ Check your baby's size and weight
  - ✓ Complete a series of play-based tests that allow medical professional to determine how well your child is developing compared to other babies his/her age.
  - ✓ Ask questions in-person about your child's feelings and behaviors. This series of question will take about 10 minutes.

#### Contact Times (Discharge and Post-discharge)

- Contact 1 at hospital discharge (of your baby)
  - ✓ Ask you to allow the medical staff to obtain your baby's weight, length, and head circumference from your baby's medical record.
  - ✓ Ask you to provide/verify your contact information
- Contact 2 by phone, home visit, or electronically at 1 month after your baby is discharged from the hospital
  - ✓ Ask you questions about how your baby is feeding, and about any urgent care/emergency room visits or hospitalizations after your baby is home. This series of questions will take about 5 minutes.
  - ✓ Ask you to provide or verify contact information
- Contact 3 by phone, home visit, or electronically when your baby is 6 months old
  - ✓ Ask you questions about how your baby is feeding, and about any urgent care/emergency room visits or hospitalizations after your baby is home. This series of questions will take about 5 minutes.
  - ✓ Ask you to provide or verify contact information
- Contact 4 by phone, home visit, or electronically when your baby is 12 months old
  - ✓ Ask you questions about how your baby is feeding, and about any urgent care/emergency room visits or hospitalizations after your baby is home. This series of questions will take about 5 minutes.
  - ✓ Ask you to provide or verify contact information

Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

- Contact 5 by phone, home visit, or electronically when your baby is 18 months old
  - ✓ Ask you questions about how your baby is feeding, and about any urgent care/emergency room visits or hospitalizations after your baby is home. This series of questions will take about 5 minutes.
  - ✓ Ask you to provide or verify contact information
- Contact 6 when your baby is 24 months old
  - ✓ Ask you to bring in your baby
    - to get his/her weight, length and head circumference
    - to have a medical professional complete a series of play-based tests that allow the medical professional to determine how well your child is developing compared to other babies his/her age.
    - Ask questions in-person about your child's feelings and behaviors. This series of question will take about 10 minutes.
  - ✓ Ask you questions about how your baby is feeding, and about any urgent care/emergency room visits or hospitalizations after your baby is home. This series of questions will take about 5 minutes.

For contact time 6, the total time needed to complete these questions and to have your baby checked by a medical professional will be about 2 to 3 hours.

#### How long will this clinical trial (study) take?

The in-hospital portion of the study will take about 1 month. The length of the hospital stay will depend on your baby's responses to treatment. Your baby's post-hospital participation in this research will take about 4 hours over the course of 2 years. There will be a total of 6 contact times. The first (at discharge) and last (when your baby is 24-months old) will be in person. The other 4 times will be either phone calls, home visits, or be done electronically. The time needed to complete these calls or electronic sessions will range from about 10 minutes to about 35 minutes. The amount of time needed for the in-person visit (contact 6) will be about 2 to 3 hours.

#### What if I say no, I do not want to be in this study?

- Nothing bad will happen.
- You/your baby can still get treatment with either morphine or methadone. Your baby's medical team will decide when the dose is changed at [insert local context here].

Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

# What happens if I say yes, but change my mind later?

- You can stop allowing your baby to be in the study at any time.
- Nothing bad will happen.
- You/your baby can still get medical care at [insert local context here].
- If you decide to stop allowing your baby to be in the study, call (*insert head researcher name*) at (*insert phone #*).

# Will it cost me anything to be in the study?

The study will not cost you anything. You or your baby's legal guardian or insurance company will be responsible for your baby's regular medical care, as usual, including the costs of the medicines and treatments used to care for your baby's NOWS symptoms.

# Will I be paid for being in the study?

Yes. We will give the person named on the signature page the following:

- 1 month post-discharge \$25.00
- Baby is 6 months old \$50.00
- Baby is 12 months old \$50.00
- Baby is 18 months old \$50.00
- Baby is 24 months old \$80.00

If you participate in all 4 of the "questionnaire-only' contact times - plus the in-person visit when the baby is 24 months old — the person named on the signature page will be paid a total of \$255.00. This is to thank the person who answered the questions for his/her time.

We will *(LOCAL CONTEXT - insert time and method of payment)*. If you change your mind and decide not to allow your baby to be in the study, the person named on the signature page will only be paid for the contact times for which he/she answered questionnaires or came for an in-person visit. The person named on the signature page will receive payment at – or near – the participation contact time.

If the person named on the signature page receives more than \$600 in one year (January-December) from *(insert local context/institution)* we may send that person a tax form, if required by law.

Informed Consent BABY ONLY Template Version #: 03

Template Date: 28-July-2021


Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

# Will being in this study help me or my baby in any way?

Being in the study may or may not help your baby. If faster weaning is successful, infants in the faster wean group will receive less morphine or methadone. The information gathered may help babies with NOWS in the future in the following ways:

- Shorten treatment time with methadone or morphine.
- Shorten hospital stays for babies.
- Decrease symptoms.
- Lower chance of return of NOWS symptoms.

# What are the risks of being in this study?

The risks are:

- Someone could find out that your baby was in the study and learn something about your baby that you did not want others to know. We will do our best to protect your/your baby's privacy.
- The questions we ask may make you feel sad or upset.
- Your baby's NOWS symptoms may return in both groups, but possibly more frequently in the fast weaning group.
- Your baby may have a harder time getting used to being home. This may be more likely if your baby is part of the fast weaning group.
- Problems among babies being treated for NOWS are not common. These problems include:
  - o seizures
  - diarrhea
  - o breathing problems
  - feeding problems
- Participation in this study does not change any need to report a newborn baby was exposed to opioid(s). Local reporting requirements for neonatal opioid exposure will be followed. These requirements are <i style="color: red;"><i style="color: red; total: reporting requirements here"></i>
- There may also be risks that are not known at this time. You will be given more information if other risks are found.

# What if I or my baby gets sick or hurt while in this study?

If your baby gets hurt when your baby is in the hospital for the study, we will help your baby get the care he/she needs. This may include first aid, emergency care, and/or follow-up care.

Template Date: 28-July-2021 
Local context version #: <insert local version #> Local context date: <insert local context date>

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

- If your baby is not here and gets hurt or sick, and think it is because of the study, do these things:
  - ✓ call your doctor or if an emergency, call 911
  - ✓ give your doctor or ER staff
    - o the name of this study, *Pragmatic, Randomized, Blinded Trial to Shorten Pharmacologic Treatment of Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)*, also called "Weaning"
    - the name of the head researcher for this study (insert researcher name)
    - o a copy of this form if you have it
  - ✓ call the head of the study (insert researcher name and 24 hour phone #)
- This treatment may be billed to you or your insurance company in the normal manner. No other form of payment is available.

# What are the alternatives to being in this study?

You do not have to allow your baby to be in this study for your baby to receive treatment for his/her condition.

If you do not want to allow your baby to be in this study, you can choose to receive the hospital's usual care for you/your baby. The hospital's usual care is treatment with either morphine or methadone and your baby's medical team will decide when the dose is changed.

#### Can my baby be taken out of the study even if I want my baby to continue?

Yes, the study doctor (or head researcher) can take your baby out of the study if:

- It is not in your baby's best interest to continue.
- Your baby has an side effect or complication related to NOWS which is considered serious and may prolong the stay in the hospital (seizure, unable to take medication by mouth either due to increased stools, breathing or feeding difficulties).
- The study is stopped for any reason.

# What information will be collected about me/my baby in the study?

During the study, we will need to learn private things about your/your baby's medical condition, including information about:

Your/your baby's background and how to contact you. Information to be collected
includes your name, address, telephone number, and other similar types of information.
You may be contacted by text, phone call, mail, home visit, or email.

Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

- ✓ If we cannot contact you from the information that you provide, we may access your/your baby's medical record to obtain contact information from your/your baby's medical record. Use of information available in the public domain may also be used to make contact.
- Information about the pregnancy of the biological mother, including physical and mental health conditions, smoking, and whether the biological mother took medications or other substances during pregnancy.
- Your baby's delivery.
- Your baby's height, weight and related measurements and information.
- Your baby's drug-test results as well as results of drug tests of the biological mother.
- Your baby's study treatment and responses to the study treatment.
- Your baby's length of time in the hospital.
- Your responses to questionnaires described in the "Description of Post-Discharge Assessment" part of this form.
- The person who is going over this consent with you can tell you exactly what information will be collected if you want to know.

#### Who will see this information? How will you keep it private?

- The local study team <insert local context, institution name> will know your name and have access to your baby's information.
- We will do our best to make sure no one outside the study knows your baby is part of the study.

To help us stay in contact with you during the study, we may ask you if you are willing to provide name(s) and contact information of back-up contact(s). It is completely up to you to decide if you want to give us additional contact information.

- ✓ If you decide to give us information for back-up contacts, you are giving us permission to contact those person(s). If we contact one of your back-ups, that person will likely find out that you are allowing your baby to be part of this study. You may also choose to provide or share other ways for us to stay in contact with you. If you agree to do provide this information, you are giving us permission to use these ways to contact you. Someone outside of the study team may then find out that you are allowing your baby to be part of this study.
- We will take your/your baby's name off of information that we collect during the study.
  - ✓ We may share your/your baby's information with your/your baby's name removed - with colleagues at the IDeA States Pediatric Clinical Trial Network Coordinating and Operations Center at University of Arkansas for Medical

Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

Sciences, the Duke Clinical Research Institute Coordinating Center, and RTI International in North Carolina.

- When we share the results of the study in meetings or medical journals, we will not include your or your baby's name or anything else that identifies you or your baby.
- There are people who make sure the study is run the right way. These people may see information from the study about you or your baby. They are:
  - ✓ NIH (National Institutes of Health), the study sponsor
  - ✓ OHRP (Office for Human Research Protections), a federal agency
  - ✓ University of Arkansas for Medical Sciences (UAMS) Institutional Review Board
  - ✓ Other institutional oversight offices
  - ✓ Investigators from other sites in the study
  - ✓ RTI International
  - ✓ FDA (Food and Drug Administration)
  - ✓ IDeA States Pediatric Clinical Trial Network Data Coordinating and Operations Center at the University of Arkansas for Medical Sciences
  - ✓ Duke Clinical Research Institute Coordinating Center
- Insert local state law requirements.

For example, state law requires that we report to the Arkansas Department of Health cases of certain diseases that a sick person could give to someone else. If we learn you have such a disease, we will share your name and contact information with the health department.

INCLUDE IF PART OF STATE LAW: State law requires we tell the authorities if we learn about possible child or adult abuse or that you might hurt yourself or someone else

#### Where and how long will my baby's information be kept?

- We will code your baby's information and keep the key to the code in a locked file or other secure location at <insert local institution>.
- Your baby's study information will also be stored, without your baby's name, at the IDeA States Pediatric Clinical Trial Network at University of Arkansas for Medical Sciences in Arkansas and at RTI International in North Carolina."
- Your baby's information will be stored indefinitely.
- Only *(insert local context, name/roles of persons)* will be able to link your baby's information to you/your baby.

Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

- Your baby's medical record will/will not indicate that your baby is participating in the study. [Statement may be change if local context requires]
- We will/will not put a copy of this consent form in your baby's medical record.

# If I/my baby stop being in the study, what will happen to any information collected from me in the study?

• We will not be able to take your baby's information out of the study after it has started.

# Will my information from the study be used for anything else, including future research?

Yes. If you allow your baby to be a participant in this study, we will keep information from this research study. The information will be de-identified (for example, a code number will be used instead of your/your child's names) so that it cannot be linked to you or your baby. The information will be placed into an appropriate NIH-approved information repository. In the future other researchers who were not part of this study may ask to use this information. Any information released to other researchers will not identify your or your baby or his/her participation in this research study.

# Will you tell me the results of the study?

• We will not notify you directly, but the results of the study will be available on a website (<a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, see below) and in medical journals. You may contact us at any time during or after the study if you have questions about the results.

#### Will you tell me anything you learn that may impact my/my baby's health?

 Yes. If we learn something about your baby that might be important for your baby's health, we will tell you.

#### What if new information comes up about the study?

- We want you to know about anything that may change your mind about allowing your baby to be in the study.
- The study team will let you know either by calling you or sending you a letter.

# Where can I find more information about this study?

A description of this study will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website any time. The ClinicalTrials.gov identifier number is NCT04214834.

Informed Consent BABY ONLY Template Version #: 03

Template Date: 28-July-2021


Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

# What if I have questions?

- Please call the head researcher of the study (insert researcher name and phone #), if you
  - ✓ have any questions about this study
  - ✓ feel your baby has been injured in any way by being in this study
- You can also call the office at UAMS that supervises research if you can't reach the study team or want to speak to someone not directly involved with this study. To do so call the UAMS Institutional Review Board (IRB) at 501-686-5667.
  - ✓ You may call the UAMS IRB if you have any questions about your baby's rights as a research participant
- [insert local context if other than researcher named above]

# By signing the document, I am saying:

- ✓ I understand that joining this study is voluntary.
- ✓ I agree to allow my baby to be in the study.
- ✓ Someone talked with me about the information in this document and answered all my questions.
- ✓ I have been asked if I wish to talk directly to the study doctor.

#### I know that:

- ✓ I can stop any and all parts of the study at any time and nothing bad will happen to me or my baby.
- ✓ I can call the office that supervises research (UAMS Institutional Review Board) at 501-686-5667 if I have any questions about the study or about my or my baby's rights.
- ✓ I do not give up any of my or my baby's rights by signing this form.
- ✓ My decision will not change my or my baby's medical care at [insert local context/site name]

.

Template Date: 28-July-2021 

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here] Institution: [insert local context here]

Sponsor: NIH Support: NIH

| I agree to allow my baby to be a participant of this stu | ıdy: |
|---|---|
| Printed Name of Parent/Guardian | |
| Signature of Parent/Guardian | Date (mm/dd/yyyy) |
| Baby's name: | |
| Relationship to baby: | |
| I agree to being contacted for future research related YES NO | to this study. |
| Printed Name of Parent/Guardian | |
| Signature of Parent/Guardian | Date (mm/dd/yyyy) |
| Is person with legal guardianship answering the quest | ions about the baby? |
| If no, the person who will be answering the questi<br>payments described in the "will I be paid" section | ` ' |
| YESNO | |
| Informed Consent BABY ONLY Template Version #: 03 Template Date: 28-July-2021 | cIRB# 260053<br> |

Template Date: 28-July-2021 Local context version #: <insert local version #> Local context date: <insert local context date>

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

| Who is the caregiver, i.e., who will receive payment for answ | wering questions about the baby? |
|---|---|
| Printed Name of Recipient | |
| Signature of Recipient | Date (mm/dd/yyyy) |
| Relationship to the baby: | |
| Name/Signature of person obtaining consent: | |
| Printed Name of Person Obtaining Consent | |
| Signature of Person Obtaining Consent | Date (mm/dd/yyyy) |

Template Date: 28-July-2021 
Local context version #: <insert local version #> Local context date: <insert local context date>

Newborns with Neonatal Opioid Withdrawal Syndrome (NOWS)

PI (researcher): [insert local context here]
Institution: [insert local context here]

Sponsor: NIH Support: NIH

# **List of Common Opioids**

# • Brand Names (generic names):

- o Demerol (meperidine)
- Dilaudid (hydromorphone)
- Lortab (hydrocodone)
- MS Contin (morphine)
- Norco (hydrocodone)
- Opana (oxymorphone)
- Oxycet (oxycodone)
- Percocet (oxycodone)
- o Zohodro ER (hydrocodone)

#### • Generic Names:

- o Buprenorphine
- o Fentanyl
- o Heroin
- Hydrocodone
- Methadone

#### • Street Names (generic names):

- o Buse, Oranges, Subs (buprenorphine)
- o Apache, China Girl, Dance Fever, Friend (fentanyl)
- o China White, Dope, H. Horse, Junk, Smack (heroin)
- Watson 387 (hydrocodone)
- o Amidone, Fizzies, Chocolate Chip Cookies (methadone)
- o M. Miss Emma, Monkey, White Stuff (morphine)
- o Hillbilly Heroin, O.C. Oxycet, Oxy (oxycodone)

Informed Consent BABY ONLY Template Version #: 03

Template Date: 28-July-2021

CIRB# 260053

